CLINICAL TRIAL: NCT02961907
Title: Pathway Taking Into Account PeriConceptional Environment for Infertile Couple
Acronym: PEPCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P140934
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2020-12

CONDITIONS: Infertility
Keywords: periconceptional habits; Pregnancy; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The usual routine course includes :
  * a clinico-biological evaluation of infertility causes
  * a laboratory staff and decision of therapeutic strategy and decision of a therapeutic strategy
  * collection of blood and sperm samples
- PEPCI group (Experimental): In the PEPCI group, the standardized assessment of the periconceptional profile is used to adapt the additional standardized intervention.
  Interventions: Procedure: PEPCI

INTERVENTIONS:
Procedure: PEPCI — Both parents will receive:
  * consultation with a psychiatrist then psychologist follow-up if required, addiction specialist physician consultation then liaison nurse follow-up if required
  * endocrinologist consultation then dietitian follow-up if required
  * actiphysician consultation and follow-up if required This program will be added to the usual routine course Both parents will receive a 3 months personalized follow-up if required from the multi disciplinary consultation and before the first ART attempt.
  Arms: PEPCI group

SUMMARY:
Infertility is defined as the inability to conceive after 12 months of unprotected intercourse, It affects approximately one in six couples pregnancy. Many lifestyle factors of the couple's pre and peri-conceptional environment (weight, diet, alcohol, tobacco, coffee, drugs, exercise, stress, sleep, pollution...) are risk factors for infertility. Weight gain, in both members of the couple, is associated with an increased risk of Assisted Reproduction Technology (ART) failure and adverse pregnancy outcome, while healthy lifestyle makes the risk of infertility three times less likely to happen. Idiopathic infertility may greatly benefit from lifestyle factors optimization.

DETAILED DESCRIPTION:
To evaluate and optimize periconceptional habits (diet and lifestyle factors) of unfertile couple may have favorable impact on conception and pregnancy.

The investigators propose to undertake a controlled trial of the efficiency of an integrated global care program. This trial of an intervention on lifestyle factors will be compared with the ""cohort multiple randomised controlled trial"" methodology in order to strengthen external validity by limiting bias that may result from initial consent to randomisation, or from deception of allocated treatment.

At any visit in a participating ART center, all attending couples will be invited to participate in an observational survey in order to allow access to their data. In this whole cohort, all eligible couples will be identified as consultations go. An ""on the fly"" randomisation process (ration 2 usual / 1 experimental) will select candidate couples from all eligible ones, who will be ten offered the experimental PEPCI intervention. In case of refusal of the experimental care, they will be given the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Couple attending a visit in an ART reproductive center (1st care regardless of the center regardless of the number of attempts in the center or in another center)
* Heterosexual infertile couple (absence of pregnancy after 12 months of unprotected intercourse)
* Men aged from 18 to 45 and women aged from 18 to 38
* Couple having not shown any opposition to the use of their data (observational study) and given their informed written consent to collect their biological samples
* Couple with good understanding of the French language
* Couple with computer equipment including webcam and internet access at home
* Affiliation to the French health insurance organism
* No-cons to the practice of adapted physical activity (non stabilized disease: diabetes, anemia, aplastic anemia, severe malnutrition, severe osteoporosis, heart or lung disease)
* Signing of the informed consent form

Exclusion Criteria:

* BMI upper 40 for one or both members of the couple
* Viral infection for one or both members of the couple (infection with HIV, Hepatitis B or C)
* Ongoing pregnancy
* One or both member of the couple medically treated for diabetes mellitus
* One or both member of the couple medically treated for a psychotic disorder
* Inability to comply with care program"
* Couple already enroll in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy will be obtained from evidence of gestational sac on ultrasound exam at 6 weeks of amenorrhea either after the first ART attempts | 3 to 12 months after the initial visit

SECONDARY OUTCOMES:
Percentage of refusal of PEPCI intervention | 12 months and 10 months additional in case of pregnancy
Assessment of patient satisfaction according Satisfaction Questionnaire (CSQ) | 12 months and 10 months additional in case of pregnancy
Assessment of impact on the health control according the Multidimensional Health Locus of Control Scale (french version) | 12 months and 10 months additional in case of pregnancy
Assessment of weight using Body mass index (BMI) expressed in units of kg/m2 | 12 months and 10 months additional in case of pregnancy
Assessment of health risk associated with excess fat around the waist using Waist Circumference WC ( measured in centimeters) | 12 months and 10 months additional in case of pregnancy
Assessment of physical activity according the International Physical Activity Questionnaire (IPAQ) | 12 months and 10 months additional in case of pregnancy
Assessment of the quality and patterns of sleep according The Pittsburgh Sleep Quality Index (PSQI) | 12 months and 10 months additional in case of pregnancy
Assessment of Anxiety and depressive disorders according Hospital Anxiety and Depression scale (HAD) | 12 months and 10 months additional in case of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Levy, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Tenon, Paris, France

REFERENCES:
- [Derived] Dupont C, Aegerter P, Foucaut AM, Reyre A, Lhuissier FJ, Bourgain M, Chabbert-Buffet N, Cedrin-Durnerin I, Selleret L, Cosson E, Levy R. Effectiveness of a therapeutic multiple-lifestyle intervention taking into account the periconceptional environment in the management of infertile couples: study design of a randomized controlled trial - the PEPCI study. BMC Pregnancy Childbirth. 2020 May 26;20(1):322. doi: 10.1186/s12884-020-2855-9. PMID 32456614